CLINICAL TRIAL: NCT00004153
Title: Sensitive RT-PCR Analysis for Melanoma Markers From Lymph Nodes and Peripheral Blood in Patients With Melanoma
Brief Title: Detection of Melanoma Markers in Lymph Nodes or Peripheral Blood of Patients With Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9308; UCCRC-9308; UCCRC-CTRC-9767; NCI-G99-1620
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Melanoma (Skin)
Keywords: stage I melanoma; stage II melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Reverse Transcriptase Polymerase Chain Reaction; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: reverse transcriptase-polymerase chain reaction
Procedure: sentinel lymph node biopsy

SUMMARY:
RATIONALE: Diagnostic procedures may improve the ability to detect the presence or recurrence of disease.

PURPOSE: Diagnostic trial to detect melanoma markers in the lymph nodes or peripheral blood of patients who have melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of performing reverse transcriptase-polymerase chain reaction (RT-PCR) for five different tumor antigen genes using lymph node samples or peripheral blood from patients with melanoma.
* Determine the ability of PCR-positive lymph nodes or peripheral blood to predict relapse of disease in these patients.
* Determine the correlation of positive PCR results from peripheral blood with disease stage.

OUTLINE: Lymph node biopsies or peripheral blood are obtained from patients. These specimens are examined by nested reverse transcriptase-polymerase chain reaction (RT-PCR) and analyzed for various tumor antigens.

Patients may choose to be told the results of this testing, but the results do not influence or change the planned therapy. Brief counseling is required to discuss the results and their potential implications.

Patients are followed for at least 2 years.

PROJECTED ACCRUAL: A total of 30 patients for the lymph node portion and 80 patients (20 per stage of disease) for the peripheral blood portion will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically proven melanoma with indication to perform sentinel lymph node biopsy or elective lymph node dissection OR
* Histologically proven or diagnosis highly suspicious for melanoma

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 50,000/mm^3
* Hemoglobin greater than 7 g/dL

Hepatic:

* PT less than 15 sec
* PTT less than 30 sec

Renal:

* Not specified

Other:

* No psychiatric illness that precludes compliance
* No other concurrent malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 1998-06; Primary Completion 2004-03 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
To determine if there is a suggestion that PCR-positive lymph nodes predict relapse of disease | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Gajewski, MD, PhD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States